CLINICAL TRIAL: NCT00462150
Title: Psychological, Physiological, and Clinical Consequences of Emotional Disclosure in Rheumatoid Arthritis (RA)
Brief Title: Effects of Home-Based Emotional Disclosure in Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NR 99-1-401
Record Dates: First submitted 2007-04-16; First posted 2007-04-18 (Estimated); Last update posted 2007-04-18 (Estimated); Status verified 2007-04

CONDITIONS: Rheumatoid Arthritis
Keywords: arthritis, rheumatoid; expressed emotion; randomized controlled trial; affect; blood sedimentation; psychophysiology; feasibility studies; intervention studies; time management
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: home-based emotional disclosure
Behavioral: time management control condition

SUMMARY:
The purpose of the study is threefold: 1) to develop a home-based emotional disclosure intervention inducing core elements of change (emotional engagement, cognitive restructuring, and positive future directedness); 2) to examine in a randomized controlled trial in patients with rheumatoid arthritis the induction of the core elements and the feasibility of the intervention for home application; and, 3) to examine the psychological, clinical, and physiological effects of the adapted emotional disclosure intervention and the modulating role of cognitive-emotional change and individual differences in emotion regulation.

DETAILED DESCRIPTION:
Emotional disclosure has been suggested to alleviate psychological and physical stress in chronically ill people. Emotional engagement, cognitive restructuring, and positive future directedness are considered core elements to induce change in emotional disclosure interventions. The aim of our randomized controlled trial in patients with rheumatoid arthritis is to examine the psychological, clinical, and physiological effects of an emotional disclosure intervention adapted for home application and the modulating role of cognitive-emotional change and individual differences in emotion regulation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of rheumatoid arthritis according to the criteria of the American College of Rheumatology (Arthritis Rheum 1988;31:315-24
* Written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2002-09; Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Depressed mood.
Cheerful mood.
Both measures at baseline, 1 week after intervention, and 3 months after intervention.

SECONDARY OUTCOMES:
Feasibility: adherence, compliance with instructions, perceived viability, clinical safety; all measured during or immediately after the intervention).
Induction of core elements: immediate negative affect change, emotion, insight, and optimism word use during the intervention.
Clinical measures: Joint score; Erythrocyte Sedimentation Rate; both measures at baseline, 1 week after intervention, and 3 months after intervention.
Physiological measures: 24-h Urinary cortisol; 24-h Urinary noradrenaline; IL-6; IFN-γ; IL-10; all measures at baseline, 1 week after intervention, and 3 months after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Henriët van Middendorp, PhD, Principal Investigator — Utrecht University, Department of Clinical and Health Psychology; Rinie Geenen, PhD, Study Chair — Utrecht University, Department of Clinical and Health Psychology; Johannes WJ Bijlsma, PhD, MD, Study Director — University Medical Center Utrecht, Department of Rheumatology & Clinical Immunology
Locations (1):
- Utrecht University, Department of Clinical and Health Psychology, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Result] van Middendorp H, Sorbi MJ, van Doornen LJ, Bijlsma JW, Geenen R. Feasibility and induced cognitive-emotional change of an emotional disclosure intervention adapted for home application. Patient Educ Couns. 2007 May;66(2):177-87. doi: 10.1016/j.pec.2006.11.009. Epub 2007 Mar 1. PMID 17336025